CLINICAL TRIAL: NCT05893225
Title: MACSiMiSE-BRAIN: Metformin add-on Clinical Study in Multiple Sclerosis to Evaluate Brain Remyelination and Neurodegeneration: a Phase II Placebo-controlled Randomized Clinical Trial
Brief Title: Metformin Add-on Clinical Study in Multiple Sclerosis to Evaluate Brain Remyelination And Neurodegeneration
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: University Hospital, Ghent (Other); Hasselt University (Other); AZ Sint-Jan AV (Other); Noorderhart Pelt (Other); National MS Center Melsbroek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MACSiMiSE-BRAIN; 2023-503190-38-00 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2022-02-28; First posted 2023-06-07 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; Primary Progressive Multiple Sclerosis; Secondary-progressive Multiple Sclerosis
Keywords: Multiple Sclerosis; Primary Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Sclerosis; Metformin; Pathologic Processes; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Brain Remyelination; Neurodegeneration
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive; Sclerosis; Pathologic Processes; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nerve Degeneration | interventions — Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): The treatment group will receive Metformin Hydrochloride oral tablets 850mg tid or bid, during a maximum of 96 weeks.
  Interventions: Drug: Metformin Hydrochloride 850 mg Oral Tablet
- Control group (Placebo Comparator): The control group will receive a matching placebo, during a maximum of 96 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin Hydrochloride 850 mg Oral Tablet — Metformin Hydrochloride oral tablets 850 mg t.i.d. or b.i.d.
  Arms: Treatment group
Drug: Placebo — Placebo matching Metformin Hydrochloride oral tablets t.i.d. or b.i.d.
  Arms: Control group

SUMMARY:
This clinical trial aims to demonstrate that metformin can prevent clinical disability in patients with progressive MS by stopping or slowing down neurodegeneration by enhancing endogenous remyelination. Patients will continue their DMT treatment: metformin or placebo will be used as add-on study treatment.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic neuroinflammatory and neurodegenerative disease leading to focal and diffuse damage of myelin sheath and axons in the central nervous system (CNS). Pathophysiologically, the adaptive and innate immune system are involved in the inflammatory process, while mitochondrial dysfunction, oxidative stress and failure of remyelination are important mechanisms leading to chronic neurodegeneration. Despite currently available disease modifying treatments (DMTs) that target the immune system, patients continue to accumulate disability. Unfortunately, no neuroprotective or remyelinating agents are available to treat progressive MS. Hence, drugs to tackle disease progression in MS represent a major unmet need. In this respect, metformin is a very interesting drug to investigate in MS patients as a neuroprotective and remyelinating therapy. Several preclinical studies in animal models of MS have shown that metformin has both anti-inflammatory, neuroprotective and remyelinating properties. A clinical study with metformin in a limited sample of MS patients did not demonstrate significant adverse events. The aim of this clinical trial is to provide evidence for the neuroprotective and remyelinating effects of metformin (I) in MS patients (P) via measurement of clinical and MRI outcome measures (O), via a multicentre randomized placebo-controlled (C) clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of non-active progressive Multiple Sclerosis (PPMS and SPMS), as evidenced by:

   1. the absence of relapses and new T2 lesions on brain MRI in the past year or longer (No Evidence of Disease Activity-2)
   2. progression of disability independent of relapses in the past 1-2 years or longer

   If progression is defined as one of the following, over the past 1-2 years or less, the patient can be included without additional review:
   * minimum increase in the EDSS of 1.0, or 0.5 from a baseline level of 2.0-5.0, and 5.5-6.0, respectively
   * ≥20% in the T25FW
   * ≥20% 9HPT
   * reduction of ≥4 points or a 10% worsening in the Symbol Digit Modality Test without concomitant depression or fatigue.

   If the investigator is in the opinion that the patient is clearly progressing, but not enough data are available to demonstrate this, a narrative needs to be provided, which will be judged by at least 2 members of the Trial Steering Committee, from a center that is not submitting the case for review.
2. Age 18-70 years inclusive
3. EDSS 2.0-6.5 inclusive
4. Able to give informed consent (signed, written) and to adhere to study procedures
5. Dutch/Flemish speaking (patient reported outcomes and questionnaires available in Dutch/Flemish)
6. Stable use of Disease Modifying Treatment (DMT) or no treatment in the past year or longer
7. Use of adequate contraceptive measures in women of childbearing potential (WOCBP)

Exclusion Criteria:

1. A medical or neurological problem other than MS that is a cause of progressive or fluctuating gait dysfunction
2. Diagnosis of diabetes mellitus or fasting glucose level of 126mg/dl or more; random glucose level of 200mg/dl or more; HbA1C of 6.5% or more at screening
3. Unable to complete T25FW
4. Unable to undergo MRI
5. Current major disease or disorder other than MS (e.g., active malignancy, significant renal insufficiency eGFR (estimated Glomerular Filtration Rate) <60 mL/min/1.73 m2, end-stage cardiopulmonary disease, alcoholism, liver insufficiency with AST (aspartate aminotransferase) >3 times Upper Limit of Normal (ULN), chronic active infection etc.) that may interfere with study procedures and/or intake of study drug
6. Pregnant or breast-feeding or planning pregnancy
7. Use of an experimental therapy in the past 6 months
8. Ongoing immune reconstitution therapy schedule (cladribine second course ended at least 12 months before inclusion, alemtuzumab second/last course at least 12 months before inclusion, Autologous Hematopoietic Stem Cell Transplantation at least 12 months before inclusion)
9. Expected change in ongoing DMT or start of DMT if untreated
10. Current use of metformin or known intolerance for metformin
11. Known sensitivity to the active substance or to any of the excipients listed in section 6.1 of the Summary of Product Characteristics.
12. All forms of acute metabolic acidosis (such as lactic acidosis, diabetic ketoacidosis), diabetic precoma.
13. Acute conditions where there is a risk of alteration of renal function, such as: dehydration, severe infection, shock occurring between screening and randomization.
14. Chronic use of NSAID

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed | From baseline to 96 weeks
  Change in walking speed as measured by the Timed 25 Foot Walk (T25FW) between baseline and 96 weeks of treatment

SECONDARY OUTCOMES:
Change in cognitive function | From baseline to 96 weeks
  Change in cognitive function as measured by Symbol Digit Modalities Test (SDMT) between baseline and 96 weeks of treatment
Change in hand function | From baseline to 96 weeks
  Change in hand function as measured by Nine-Hole Peg Test (9HPT) between baseline and 96 weeks of treatment
Change in EDSS | From baseline to 96 weeks
  Change in Expanded Disability Status Scale. The EDSS is a disability scale that ranges in 0.5-point steps from 0 (normal) to 10.0 (death) and is determined based on functional system scores (FSS) that are assigned after a standardized clinical neurological examination.
Change in brain volume | From baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
  Change in brain volume (whole brain volume and gray matter volume) from baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
Change in T2 lesion volume | From baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
  Change in T2 lesion volume from baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
Change in T1 lesion volume | From baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
  Change in T1 lesion volume from baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
Change in brain magnetic resonance imaging diffusion tensor imaging (MRI-DTI) metrics | From baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
  Change in brain MRI-DTI metrics from baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks

OTHER OUTCOMES:
Change in quality of life measured by EQ-5D-5L | From baseline to 96 weeks
  Change in quality of life as measured by EuroQol 5-dimension, 5-level (EQ-5D-5L) questionnaire between baseline and 96 weeks of treatment. The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This tool also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable.
Change in quality of life measured by MSIS-29 | From baseline to 96 weeks
  Change in quality of life as measured by Multiple Sclerosis Impact Scale-29 between baseline and 96 weeks of treatment. The MSIS, is a 29-item patient-reported measure of the physical and psychological impacts of MS. Patients are asked to rate how much their functioning and well-being has been impacted over the past 14 days on a 4-point scale, from "Not at all" (1) to "Extremely" (4).
Change in the Composite endpoint | From baseline to 96 weeks
  Change in the Composite endpoint as measured by Overall Disability Response Score (ODRS) between baseline and 96 weeks of treatment. The ODRS is based on changes in EDSS, T25FW and 9HPT. At each time point, in individual patients, the scores of the four components are summed, which leads to a total score ranging from +4 to -4. A positive ODRS score means that there is a disability improvement compared to baseline and a negative ODRS score means a disability worsening from baseline.
Change in 2 minute walk test | From baseline to 96 weeks
  Change in 2 minute walk test between baseline and 96 weeks of treatment
Change in number of susceptibility weighted imaging (SWI) lesions | From baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
  Change in number of SWI lesions from baseline to 48 weeks, from baseline to 96 weeks and from 48 to 96 weeks
Change in caregiver strain index (CSI) | From baseline to 96 weeks
  Change in caregiver strain index from baseline to 96 weeks. It is a 13-question tool that measures strain related to care provision. There is at least one item for each of the following major domains: Employment, Financial, Physical, Social and Time.
Health resource questionnaire | From baseline to 96 weeks
  This questionnaire is adapted from Kobelt et al. and will be used to generate data for health economic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Willekens, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (5):
- Belgium (5):
  - AZ Sint-Jan Brugge, Bruges
  - Antwerp University Hospital, Edegem
  - University Hospital Ghent, Ghent
  - National MS Center Melsbroek, Melsbroek
  - Noorderhart, Overpelt

IPD SHARING:
Plan to Share IPD: Yes
Protocol section 14.9 Access to the Study Data describes this in detail.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After peer-reviewed publication of study protocol and clinical trial results
Access Criteria: See protocol section 14.9 Access to the Study Data

REFERENCES:
- [Background] De Keersmaecker AV, Van Doninck E, Popescu V, Willem L, Cambron M, Laureys G, D' Haeseleer M, Bjerke M, Roelant E, Lemmerling M, D'hooghe MB, Derdelinckx J, Reynders T, Willekens B. A metformin add-on clinical study in multiple sclerosis to evaluate brain remyelination and neurodegeneration (MACSiMiSE-BRAIN): study protocol for a multi-center randomized placebo controlled clinical trial. Front Immunol. 2024 Feb 21;15:1362629. doi: 10.3389/fimmu.2024.1362629. eCollection 2024. PMID 38680485